CLINICAL TRIAL: NCT02686489
Title: Large Volume Nebulizers Versus Heated Humidity in Spontaneously Breathing Tracheostomy Patients
Brief Title: Humidity Therapy for Spontaneously Breathing Tracheostomy Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll enough subjects to answer the research questions
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16010603
Record Dates: First submitted 2016-02-04; First posted 2016-02-19 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heated humidification (HH) (Experimental): Addition of water vapor (molecular water) to the inspired gas of spontaneously breathing tracheostomy patients.
  Interventions: Other: Heated humidification
- Cool bland aerosol (LVN) (Active Comparator): Addition of particulate water to the inspired gas of spontaneously breathing tracheostomy patients.
  Interventions: Other: Cool bland aerosol

INTERVENTIONS:
Other: Heated humidification — Water vapor (molecular water) will be added to the inspired gas of the spontaneously breathing tracheostomy patient by using the Fisher & Paykel Healthcare, (Auckland, New Zealand) AIRVO 2 Humidification System. The AIRVO 2 will provide respiratory gas flow at 2-60 L/min) that is conditioned to 37° C, 34° C, or 31° C (based on patient comfort) and 100% relative humidity via a heated breathing circuit.
  Arms: Heated humidification (HH)
Other: Cool bland aerosol — Aerosol (particles of water suspended in gas) generated by a flow of gas through a pneumatically powered large volume jet nebulizer filled with sterile water (for inhalation) attached to a gas source via a flowmeter set between 10-15 L/min will add moisture to the inspired gas of the spontaneously breathing tracheostomy patient. The cold bland aerosol set-up will consist of corrugated aerosol tubing with one end connected to the nebulizer output port and the other end connected to a tracheostomy mask.
  Arms: Cool bland aerosol (LVN)

SUMMARY:
The goal of the study is to compare the safety and efficacy of molecular water and bland aerosol therapy (particulate water) in providing adequate humidity to the inspired gas of spontaneously breathing tracheostomy patients.

DETAILED DESCRIPTION:
Currently, there is no empirical evidence of the significant superior efficacy of particulate water via large volume nebulizer (LVN), in providing humidity therapy to spontaneously breathing tracheostomy patients over molecular water via heated humidifier. Large volume nebulizers are a commonly used therapy in clinical practice for tracheostomy patients. However, in terms of an optimal modality for providing humidification when the upper-airway is bypassed, there is much controversy. Much of the available literature has looked into a comparison between heated humidity (HH) and heat and moisture exchangers (HMEs) in intubated patients in crossover studies and case studies. In addition, they have seen overall greater outcomes in HH. Nonetheless, no recent studies have directly compared the use of HH and LVNs during humidity therapy in spontaneously breathing tracheostomy patients. Although a couple of past studies have directly compared the two humidity types in spontaneously breathing patients with a bypassed upper airway, no research has been conducted as follow-up to these past studies. Furthermore, these studies were restricted to outcomes of arterial oxygenation and also had limitations due to the short duration of the studies and small sample sizes.

A tracheostomy is an artificial airway characterized by a surgically made incision that passes through the anterior neck and into the trachea. A tube is placed inside the hole created by the incision to provide a patent airway for an individual with impaired respiratory function to breathe. Approximately 100,000 tracheostomy procedures are performed annually in the United States. The burden of cost for tracheostomy patients in the United States related to the duration of hospital stay for these patients is a major factor that has contributed to the resurgence of interest in the management of tracheostomy patients. According to data from the Agency for Healthcare Research and Quality (AHRQ), in 2009, the average length of hospital stay for a tracheostomy patient was 29 days. In 2013, an analysis of data on patients with acute respiratory failure from 90% of the non-profit academic medical centers in the United States revealed high resource utilization and high morbidity rates for tracheostomy patients. The analysis also revealed that tracheostomy patients with acute respiratory failure had on average, a longer intensive care unit stay (24.3 days) than non-tracheostomy patients with acute respiratory failure (6.6 days). Mean hospital stay was also higher for tracheostomy patients (36.6 days) than non-tracheostomy patients (11.3 days). Moreover, on average, the total hospital cost for tracheostomy patients was $285,509 and $ 86,118 for non-tracheostomy patients.

Management of a tracheostomy is a complex undertaking and includes many components that span several healthcare disciplines, including tube and stoma care, humidity therapy, communication and swallowing strategies, emergency management, and weaning and decannulation. In recent years, clinicians worldwide have demonstrated a renewed interest in the management of tracheostomy patients due to recognition of preventable adverse outcomes for many of these patients. The United Kingdom's 2014 report by the National Confidential Enquiry into Patient Outcome and Death (NCEPOD) on the care received by tracheostomy patients concluded that tracheostomy management is suboptimal. Since tracheostomy management is a complex, multi-disciplinary endeavor, recent research has advocated the use of a multidisciplinary tracheostomy team. One notable collective is the Global Tracheostomy Collaborative; this collaboration consists of a multidisciplinary team of physicians, nurses, respiratory therapists, speech therapists, and patients working together to find best practices and improve the clinical outcomes centered on tracheostomy care. As part of their mission, they state that, "through multidisciplinary care, a standardization of care, broad staff educations, and patient and family involvement, these critical key drivers serve to continue to bring about improvements in tracheostomy care." In an effort to improve the care of tracheostomy patients, an expert panel convened by the American Academy of Otolaryngology - Head and Neck Surgery developed a Clinical Consensus Statement on the management of these patients. The authors of the consensus statement noted that current approaches to tracheostomy care are inconsistent among clinicians and between different institutions. Consequently, the primary goal of the consensus statement is to reduce variances in clinical practice when managing tracheostomy patients, and minimizing complications. Aspects of tracheostomy management that are addressed by the clinical consensus statement include initial tube change, management of emergencies and complications, decannulation protocol, management of tube cuffs and communication devices, and specific patient and caregiver needs. With regard to humidification, the expert panel reached the following consensus: (i) humidification should be used during the immediate postoperative period and as necessary thereafter, (ii) humidification should be used if a patient requires mechanical ventilation, and (iii) humidification should be used for patients with a history of thick secretions.

Inadequate humidification for tracheostomized patients can result in an assortment of adverse complications, which ultimately negatively impact the epithelial integrity of the airway. This is the case in situations where patients breathe the cold, dry air delivered by the gas supply systems of hospitals. According to the American Association for Respiratory Care (AARC) clinical practice guidelines for humidification, adequate humidification requirements when the upper airway is bypassed entails a humidity output of 33-44 mg H2O/L, with a 100% relative humidity at 34-41°C. Several types of devices may be used in the clinical setting to provide humidity therapy. Thus, awareness of the type of humidity therapy they provide is just as important as understanding their principles of operation, application, as well as their potential hazards. The use of large volume jet nebulizers (LVNs) is very common in respiratory care practice as a modality for humidification therapy. These devices are pneumatically powered, and deliver cool/bland aerosol by using a variable oxygen diluter and water passing through a jet nozzle. The aerosols provided by LVNs are usually unheated, cool and bland. Thus, one would expect to see complications arise from the wide use of LVNs in the clinical setting. However, superior efficacy of a device still remains questionable and as evident, there exists huge inadequacies in studies on humidification of spontaneously breathing tracheostomy patients and overall tracheostomy care. Heated humidifiers entail the use of active humidity, which use energy and water external to the body (e.g. a wick humidifier or passover humidifier) for conditioning inspired gases. Passive heated humidifiers on the other hand, rely on body temperature and the humidity gradient between the body and external environment. One of the most widely used types of passive humidifiers is the heat and moisture exchanger (HME), which contains a condenser element designed to enhance capturing the exhaled moisture (in the form of water vapor) from the patient's breath, then transfer and release this moisture back into the inspired air on the next breath.

Kuo et al. compared bland aerosol and heated humidity in spontaneously breathing patients with nasal endotracheal tubes and normal lungs and found a detrimental effect on patient's oxygenation status when using a heated jet nebulizer for short-term use. It is interesting to note that these effects were improved by exchanging therapy to heated humidity. However, contradictory results were observed by Rozsasi et, al. in which tracheal humidity remained at higher levels after use of particulate aerosol spray (300µL H2O/L air at 26°C, 90% relative humidity) in comparison to molecular water vapor (32µL H2O/L air at 32°C, 100% relative humidity). Studies have in addition compared the use of heat and moisture exchangers (HMEs), a type of passive humidification, in comparison to HH in mechanically ventilated patients and have shown mixed results regarding the superior efficacy of one over the other. However, a recent systematic review found no difference in adverse clinical events such as artificial airway occlusion, mortality, pneumonia, or respiratory complications between HH and HME.

The goal of the proposed study is to help bridge the knowledge gap regarding the management of patients with tracheostomy tubes and to improve patient care by contributing to the development of clinical practice guidelines relevant to humidity therapy for spontaneously breathing tracheostomy patients.

Methodology Study Design and Population The proposed study will be conducted at Rush University Medical Center (RUMC) in Chicago, Illinois. Using the medical center's electronic medical database (Epic), a current list of tracheostomy patients will be acquired as the accessible population. From this patient list, a sample of those that fit the inclusion and exclusion criteria will be used as the study sample. Patients from the intensive care unit (ICU) as well as various acute care floors will be included in the study. Participants will be approached individually to request consent for participation in the proposed study, and their cooperation will be emphasized as being strictly voluntary.

Consecutive sampling will be employed as the sampling technique to include every available tracheostomy patient who meets the inclusion criteria, in order to attain results as close to the target population of spontaneously breathing tracheostomy patients as possible. This is the most robust nonprobability sampling strategy because since the complete accessible population is studied, the chance of observing a representative subset of the population is increased.

Using the design of a prospective randomized control trial (RCT), patients will be randomly assigned to either of two groups: (A) humidity therapy with aerosol using a large volume nebulizer, or (B) humidity therapy with molecular water vapor using heated humidity. A sample size greater than 100 participants will be the target, as the proposed study intends to address the small sample size limitations of previous studies. Furthermore, the study period of approximately 60 days is desired to observe the long-term outcomes that may result.

ELIGIBILITY:
Inclusion Criteria

* Greater than eighteen years old
* Tracheotomized less than or equal to two weeks before entry into the study
* Spontaneously breathing

Exclusion Criteria

* Less than eighteen years old
* Tracheotomy performed more than two weeks prior to enrolment in the study
* Mechanically ventilated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-08-11 (Actual)

PRIMARY OUTCOMES:
Clinical pulmonary infection score (CPIS) | Within the first 7 days of initiation of the intervention
  Pulmonary infection rate as determined by CPIS score

SECONDARY OUTCOMES:
Incidences of tracheostomy tube occlusion with respiratory secretions (mucus plugging of tracheostomy tube) | Within the first 7 days of initiation of the intervention
  Any incidence of tracheostomy tube occlusion observed during the first 7 days of the intervention
Pulmonary complications | Within the first 7 days of initiation of the intervention
  Incidences of bronchospasm, atelectasis, hospital acquired pneumonia (HAP), ICU re-admission, and respiratory failure requiring mechanical ventilation
Cost of care | Within 3 months of the study's completion date
  defined as the overall hospital costs between patients using a specific type of humidity therapy (LVN/HH) from the beginning of the study to the end of the study
Length of hospital stay | Within 3 months of the study's completion date
  Duration of stay in the hospital by the tracheostomy patient from the initiation of the study to the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards EA, Byrnes CA. Humidification difficulties in two tracheostomized children. Anaesth Intensive Care. 1999 Dec;27(6):656-8. doi: 10.1177/0310057X9902700618. PMID 10631425
- [Background] McNamara DG, Asher MI, Rubin BK, Stewart A, Byrnes CA. Heated humidification improves clinical outcomes, compared to a heat and moisture exchanger in children with tracheostomies. Respir Care. 2014 Jan;59(1):46-53. doi: 10.4187/respcare.02214. Epub 2013 Jun 13. PMID 23764867
- [Background] Kuo CD, Lin SE, Wang JH. Aerosol, humidity and oxygenation. Chest. 1991 Jun;99(6):1352-6. doi: 10.1378/chest.99.6.1352. PMID 2036815
- [Background] Rozsasi A, Durr J, Leiacker R, Keck T. Delivery of molecular versus particulate water in spontaneously breathing tracheotomized patients. Head Neck. 2007 Jan;29(1):52-7. doi: 10.1002/hed.20473. PMID 16983692
- [Background] Kacmarek, Robert, James Stoller, Albert Heuer. Egan's Fundamentals of Respiratory Care, 10th Edition. Mosby, 2013. VitalBook file.
- [Background] Williams R, Rankin N, Smith T, Galler D, Seakins P. Relationship between the humidity and temperature of inspired gas and the function of the airway mucosa. Crit Care Med. 1996 Nov;24(11):1920-9. doi: 10.1097/00003246-199611000-00025. PMID 8917046
- [Background] The Global Tracheostomy Collaborative. Tracheostomy 101. Retrieved 12/15/2015 at http://globaltrach.org/tracheostomy.
- [Background] Yu M. Tracheostomy patients on the ward: multiple benefits from a multidisciplinary team? Crit Care. 2010;14(1):109. doi: 10.1186/cc8218. Epub 2010 Jan 29. PMID 20156313
- [Background] Agency for Healthcare Research and Quality (AHRQ), HCUP-net National and regional estimates on hospital use for all patients from the HCUP Nationwide Inpatient Sample (NIS), 2009.
- [Background] Freeman BD, Stwalley D, Lambert D, Edler J, Morris PE, Medvedev S, Hohmann SF, Kymes SM. High resource utilization does not affect mortality in acute respiratory failure patients managed with tracheostomy. Respir Care. 2013 Nov;58(11):1863-72. doi: 10.4187/respcare.02359. Epub 2013 Apr 30. PMID 23650434
- [Background] Wilkinson KA, Freeth H, Martin IC. Are we 'on the right trach?' The National Confidential Enquiry into Patient Outcome and Death examines tracheostomy care. J Laryngol Otol. 2015 Mar;129(3):212-6. doi: 10.1017/S0022215115000158. Epub 2015 Feb 3. PMID 25645673
- [Background] Mitchell RB, Hussey HM, Setzen G, Jacobs IN, Nussenbaum B, Dawson C, Brown CA 3rd, Brandt C, Deakins K, Hartnick C, Merati A. Clinical consensus statement: tracheostomy care. Otolaryngol Head Neck Surg. 2013 Jan;148(1):6-20. doi: 10.1177/0194599812460376. Epub 2012 Sep 18. PMID 22990518
- [Background] Cetto R, Arora A, Hettige R, Nel M, Benjamin L, Gomez CM, Oldfield WL, Narula AA. Improving tracheostomy care: a prospective study of the multidisciplinary approach. Clin Otolaryngol. 2011 Oct;36(5):482-8. doi: 10.1111/j.1749-4486.2011.02379.x. PMID 21838807
- [Background] Volsko, Teresa A., Robert L. Chatburn, and Mohamad F. El-Khatib.
- [Background] American Association for Respiratory Care; Restrepo RD, Walsh BK. Humidification during invasive and noninvasive mechanical ventilation: 2012. Respir Care. 2012 May;57(5):782-8. doi: 10.4187/respcare.01766. PMID 22546299
- [Background] Branson RD, Davis K Jr, Campbell RS, Johnson DJ, Porembka DT. Humidification in the intensive care unit. Prospective study of a new protocol utilizing heated humidification and a hygroscopic condenser humidifier. Chest. 1993 Dec;104(6):1800-5. doi: 10.1378/chest.104.6.1800. PMID 8252968
- [Background] Kelly M, Gillies D, Todd DA, Lockwood C. Heated humidification versus heat and moisture exchangers for ventilated adults and children. Cochrane Database Syst Rev. 2010 Apr 14;(4):CD004711. doi: 10.1002/14651858.CD004711.pub2. PMID 20393939